CLINICAL TRIAL: NCT01157403
Title: Autologous Transplantation of Mesenchymal Stem Cells for Treatment of Patients With Onset of Type 1 Diabetes
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lu Debin (Other)
Responsible Party: Sponsor-Investigator, Lu Debin, Southwest Hospital, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ldb201001
Record Dates: First submitted 2010-07-02; First posted 2010-07-07 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Evidence of Liver Transplantation
Keywords: mesenchymal stem cells
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cells (Experimental): To study the safety and efficacy of autologous transplantation of bone marrow mesenchymal stem cells in treatment of newly diagnosed patients with T1DM.
  Interventions: Biological: Autologous transplantation

INTERVENTIONS:
Biological: Autologous transplantation — Autologous transplantation of bone marrow mesenchymal stem cells (approximately 2.5 x 106 cells/kg body weight) intravenously
  Other Names: SWH2010A19

SUMMARY:
Type 1 diabetes mellitus (T1DM)is characterized by the autoimmune destruction of the pancreatic β cells; as a result, patients with T1DM are dependent on exogenous insulin to control their blood glucose continuously. Bone marrow-derived mesenchymal stem cells has been shown in many animal studies their potential cure for T1DM,which could not only address the need for β-cell replacement but also control of the autoimmune response to cells which express insulin. Therefore it is need to study the safety and efficacy of autologous bone marrow mesenchymal stem cells in treatment of newly diagnosed patients with T1DM.

DETAILED DESCRIPTION:
Autologous transplantation of Bone marrow mesenchymal stem cells(approximately 2.5 x 106 cells/kg body weight) intravenously

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent from patients or Child guardian
2. Confirmed diagnosis of type 1 diabetes by ADA criteria less than 18 weeks •

Exclusion Criteria:

1. Body Mass Index >30
2. Presence of acute stage as Active infection,recent myocardial infarction, recent cerebral vascular accident (CVA) or acute renal failure.
3. Severe Organ damage(e.g. lung disease, or hematopoietic dysfunction, or liver dysfunction).
4. Infectious diseases, e.g. HIV infection, or hepatitis B or C infection
5. Presence of malignancy

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
C peptide release test | 6 Months after intervention
  The concentration of c-peptide at 90 minutes after the start of the C-peptide release test at 24 Months following the infusion or not with bone marrow mesenchymal stem cells

CONTACTS AND LOCATIONS:
Overall Officials: chen bing, doctor, Study Director — Endocrine Department, the south west Hospital of the Third Military Medical University
Locations (1):
- Endocrine Department, the south west Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality, China